CLINICAL TRIAL: NCT02537639
Title: Impact of Simulator-based Training in Transoesophageal Echocardiography
Acronym: ISITOE
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Andreas Bloch
Record Dates: First submitted 2015-07-29; First posted 2015-09-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Imaging of Heart Disease
Keywords: Simulator in transesophageal echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Control group. Standard teaching in transesophageal echocardiography.
- Intervention group: Intervention group. Additional teaching with a transesophageal echocardiography simulator.
  Interventions: Device: Transesophageal echocardiography simulator

INTERVENTIONS:
Device: Transesophageal echocardiography simulator
  Groups: Intervention group

SUMMARY:
The investigators would like to evaluate how well intensive care trainees without previous experience in transesophageal echocardiography are able to perform a transesophageal echocardiography study in the clinical setting after completing a simulator based training compared to conventional training.

DETAILED DESCRIPTION:
Background

Echocardiography is currently the sole imaging modality at the bedside that provides real-time information on cardiac anatomy and function. Echocardiography is increasingly used in the intensive care unit (ICU) setting for the focussed hemodynamic assessment of patients with cardiorespiratory compromise. The principal role for focussed echocardiography is the time-sensitive assessment of the symptomatic patient. This evaluation primarily includes the assessment for pericardial effusion, the evaluation of relative chamber size, global cardiac and valvular function and patient volume status. The clinical impact of echocardiography for the treatment of critically ill patients with hemodynamic compromise is well documented and increasing general consensus exists, that all physicians in charge of critically ill patients should be trained in focussed echocardiography. Accordingly there is an urgent need for specific training in echocardiography.

Transoesophageal echocardiography (TOE) is besides transthoracic echocardiography (TTE) the main imaging modality in the ICU setting. TTE image quality is often compromised by lung inflation in ventilated patients or by the presence of dressings or drains in locations used for image acquisition. It thus seems reasonable to suggest that every critical care physician should be able to perform a focused TOE. However, a multitude of barriers continue to limit TOE training including time constraints in busy ICUs, limited number of appropriate cases and a lack of experienced teaching faculty. Proficiency in TOE image acquisition requires in-depth knowledge of three-dimensional cardiac anatomy and repetitive supervised hands-on experience to develop the necessary manual skills. Typically TOE skill acquisition occurs in real time in the ICU while caring for a patient, thus the time that can be devoted to training is limited. However, using a semi-invasive imaging modality in ICU patients for training solely for training purposes is problematic due to the associated (minimal) risks and patient discomfort. Recently commercially available TOE simulation systems have been introduced. These systems allow for patient-independent training of TOE skills using simulations of the human heart. When used as an educational adjunct standardized TOE simulation training in a virtual reality environment may lead to a more rapid development of psychomotor skills. TOE simulators also offer the possibility to simulate pathological conditions of the heart and thus may facilitate training in image interpretation.

The purpose of this study is to determine the effectiveness of a simulator based TOE training curriculum to train all necessary components of focused critical care echocardiography in accordance with the basic perioperative transesophageal examination as defined by the American Society of Echocardiography and the Society of Cardiovascular Anesthesiologists. This includes the psychomotor skills necessary for obtaining echocardiographic images of sufficient quality according to established quality scoring systems and the ability of recognizing the relevant anatomic structures as well as image interpretation when evaluating a hemodynamically compromised patient.

Objective

To evaluate the effect of a simulator in the training for transesophageal echocardiography

Methods

The investigators will perform a prospective, observational trial investigating the impact of simulator TOE training in novice operators on quality of imaging, correct image interpretation and resource use when performing a focussed TOE examination in ICU patients. Forty-fife ICU trainees without previous hands-on echocardiography skills will undergo a formal training consisting of 4 hours of theoretical instructions including basics of transesophageal echocardiography, cardiac anatomy, standard views as well as physiology and pathophysiology. Instructions will be provided by expert TOE operators. 30 of these trainees will additionally be trained using the HeartWorks TOE simulator. This training consists of 4 sessions of supervised practice using the TOE simulator.

After conclusion of the training program the trainees will perform one basic perioperative echocardiography study using the HeartWorks TOE simulator and two basic perioperative echocardiography studies in real ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* No prior hands-on training in echocardiography
* Trainee in critical care
* Written informed consent

Exclusion Criteria

* Prior hands-on training in echocardiography

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trainees in critical care
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Quality of acquired images | After training completion, expected to be on average between 1 and no more than 5 days
  Assessed by two cardiologists based on predefined quality criteria

SECONDARY OUTCOMES:
Time needed to perform the examination | After training completion, expected to be on average between 1 and no more than 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bloch, Principal Investigator — Department for critical care, university hospital bern
Locations (1):
- Department for Critical Care, Bern, Switzerland

REFERENCES:
- [Derived] Bloch A, von Arx R, Etter R, Berger D, Kaiser H, Lenz A, Merz TM. Impact of Simulator-Based Training in Focused Transesophageal Echocardiography: A Randomized Controlled Trial. Anesth Analg. 2017 Oct;125(4):1140-1148. doi: 10.1213/ANE.0000000000002351. PMID 28817424